CLINICAL TRIAL: NCT04780425
Title: A Randomised Parallel-group Multi-centre Study to Evaluate the Effect of Structured Diabetes Self-management Education Versus Standard of Care on Glycaemic Control, Self-efficacy and Quality of Life in Adults in Two Low Resource Settings in Accra Subsequent to COVID-19
Brief Title: Structured Diabetes Self-Management Education and Care Outcomes in Adults liVIng With Type 2 Diabetes in Accra, Ghana
Acronym: SMSCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korle-Bu Teaching Hospital, Accra, Ghana (Other)
Collaborators: University of Leicester (Other); Utrecht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KBTH-IRB 100017512020
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: structured diabetes self-management education; DESMOND; SSA
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Persons delivering the intervention are not involved in patient care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DESMOND (Experimental): receive usual care plus a structured diabetes self-management education program delivered once over 6hours
  Interventions: Behavioral: DESMOND
- USUAL CARE (Active Comparator): Receive usual care as per standard treatment guidelines of ghana unstructured education during clinic visits for routine care
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: DESMOND — as previously described
  Arms: DESMOND
Other: usual care — usual care as per standard treatment guidelines of Ghana unstructured/adhoc diabetes education during clinic visits
  Arms: USUAL CARE

SUMMARY:
We aim to study the effect of a structured diabetes education program (DESMOND) on diabetes outcomes in a ghanaian population over 3 months

DETAILED DESCRIPTION:
Protocol summary Background: Health systems in low-income countries are overburdened. Corona virus disease-19 (COVID-19) is a pandemic caused by a novel corona virus, Severe acute respiratory syndrome-corona virus 2 (SARS-CoV2) while diabetes is a long-standing global epidemic. COVID-19 further stresses the already overburdened health systems and Public Health measures to contain COVID-19 have severely disrupted health service delivery, particularly routine care. Delivery of diabetes specific education has traditionally been tied to routine visits and delivered in-person. COVID-19 will likely continue to influence service delivery beyond the pandemic, thus alternative ways of delivering diabetes specific education is needed.

Diabetes self-management education is vital to providing diabetes care. It equips patients with critical knowledge and skills for self-care. Recent edicts to stay home in relation to COVID-19 have further heightened the importance of self-care. Appropriate self-management behaviours are associated with lower levels of diabetes related distress, better quality of life and diabetes outcomes overall. Maintaining tight glycaemic control, early in diabetes is associated with fewer microvascular complications and vice versa. Complications of diabetes are prevalent in low resource settings in Africa; partly because of inadequate knowledge on self-care. Diabetes self-management education which is structured and tailor-made for low resource settings may modify self-care behaviors and result in improved self-care, glycaemic control and quality of life.

Aim:

To compare structured diabetes self-management education with standard of care among adults living with type 2 diabetes

Methods:

A prospective parallel-group randomised controlled trial with three months follow-up will be conducted in KBTH Polyclinic/Family Medicine Centre and Weija Gbawe Municipal Hospital, two primary care facilities in Accra. Participants will be individually randomised to standard of care or 6 hours of structured diabetes self-management education (DSME) delivered in person on one day . Each arm will have hundred participants. The standard of care arm will receive unstructured DSME as per existing protocols at each study site. The study population will be adults living with diabetes. The primary outcome, mean glycated haemoglobin (HbA1c ) will be measured at three months.

Expected outcomes:

It is expected that there will be no difference in change in mean glycaemic control, self-efficacy or quality of life at three months between the two arms.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria

1. Self-identified as Ghanaian
2. Ability to speak either English and or Twi
3. be aged > 18 years
4. be receiving treatment at the study site as an out-patient
5. be willing to accept the 6-hour DSME intervention
6. be physically able to participate
7. be primarily responsible for their own care
8. be ambulant at time of recruitment
9. be able to participate in activities in a group setting
10. have permanent residence in Greater Accra

Exclusion Criteria:

1. known to have cognitive defects
2. known to have type I diabetes
3. known to be pregnant at the time of recruitment or planning to become pregnant during the study or have given birth less than three months prior to recruitment
4. known to have sickle cell disease
5. Participating in another intervention study at time of recruitment
6. known to have chronic medical complications of diabetes (cardiac, renal, neuropathy, hepatic) or systemic illness at the time of recruitment
7. recruitment of a member of the patients household for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Change in mean glaciated heamoglobin (HbA1c) at three months | 3 months
  change in glycaemic control

SECONDARY OUTCOMES:
Change in mean fasting plasma glucose (FPG) at three months | 3 months
  change in fasting plasma glucose
Change in mean fasting blood glucose (FBG) at three months | 3 months
  change in fasting blood glucose
Change in mean blood pressure (BP) at three months | 3 months
  change in blood pressure
Change in waist circumference (WC) at three months | 3 months
  change in waist circumference
Change in neck circumference (NC) at three months | 3 months
  change in neck circumference
Change in body weight (BW) at three months | 3 months
  change in body weight
Change in problem areas in diabetes (PAID-5) scores | 3 months
  Change in diabetes related distress at three months, scored from 0 to 4 for each question. minimum score is 0 maximum score is 20, higher scores mean better outcomes
Change in mean summary of diabetes self-care activities (SDSCA) score at three months | 3 months
  change in self-efficacy, min score 0 and max score 7 for each question, higher scores mean better outcomes
Change in mean WHO quality of life (WHOQoL BREF) score at three months | 3 months
  change in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Lamptey, FWACP; MSc, Principal Investigator — Korle Bu Teaching Hospital
Locations (2):
- Ghana (2):
  - Korle Bu Teaching Hospital, Accra
  - Weija Gbawe Municipal Hospital, Accra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamptey R, Amoakoh-Coleman M, Barker MM, Iddi S, Hadjiconstantinou M, Davies M, Darko D, Agyepong I, Acheampong F, Commey M, Yawson A, Grobbee DE, Adjei GO, Klipstein-Grobusch K. Change in glycaemic control with structured diabetes self-management education in urban low-resource settings: multicentre randomised trial of effectiveness. BMC Health Serv Res. 2023 Feb 24;23(1):199. doi: 10.1186/s12913-023-09188-y. PMID 36829179